CLINICAL TRIAL: NCT06718868
Title: Evaluation of the Effect of Pectoral Nerve Block II on Acute and Chronic Pain in Patients Undergoing Oncological Breast Surgery
Status: Completed | Type: Observational
Sponsor: Irem Erkan (Other)
Responsible Party: Sponsor-Investigator, Irem Erkan, Resident Doctor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Organization: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Other Study IDs: E-48670771-514.99-232052317
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Breast Carcinoma; Chronic Pain
Keywords: Oncological breast surgery, PECS II Block, chronic pain, acute pain
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain; Acute Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Patients in Group 1 were defined as those who received PECSII Block in addition to intravenous analgesia.
- Group 2: Patients in Group 2 were defined as patients who received intravenous analgesia only.

SUMMARY:
The aim of this observational study is to evaluate the effect of Pectoral Nerve Block II (PECSII) on the development of pain in the acute and chronic periods in female patients over the age of 18 who underwent oncological breast surgery. The main questions it aims to answer are:

Is PECSII blockade applied to patients undergoing oncological breast surgery effective on acute pain scores compared to the non-blockade group? Is there a difference between the group with block and the group without block in terms of the development of chronic pain in the evaluation made at the 3rd month after surgery? The analgesia method applied to the patients will be recorded in the patient files and acute and chronic pain scores will be evaluated. Chronic pain score evaluation will be made by telephone survey.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be operated under general anesthesia
* ASA score I-II-III patients
* Non-pregnant patients
* Patients who agreed to participate in the study

Exclusion Criteria:

* Patients with coagulopathy
* Patients who underwent bilateral mastectomy
* Patients with chest wall anomalies
* Patients with neuropathic pain before surgery
* Patients who did not agree to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 128 patients who met the inclusion criteria were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of PECSII block on the development of chronic pain in patients undergoing oncological breast surgery | 3 months
  Female patients over 18 years of age, non-pregnant, cooperative, and who agreed to participate in the study, who underwent oncological breast surgery, were contacted by phone in the 3rd month post-operation and evaluated for the development of chronic pain using the PAIN Detect pain scale.Only patients who received routine intravenous analgesia and patients who received PECSII block in addition to routine intravenous analgesia were included in the study. The patients were divided into two groups. The development of chronic pain in the block group was compared with the patients in the non-block group. The surgical technique applied to the patients was recorded from the patient files. The relationship between surgical technique and pain occurrence was evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Serap Karacalar, Prof., Study Director — Prof. Dr. Cemil Tascioglu Education and Research Hospital; İrem Erkan, M.D., Principal Investigator — Prof. Dr. Cemil Tascioglu Education and Research Hospital
Locations (1):
- Prof. Dr. Cemil Tascıoglu Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided